CLINICAL TRIAL: NCT00249626
Title: Therapists to Administer Contingency Management-Therapist Phase
Brief Title: Therapists to Administer Contingency Management-Therapist Phase - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: NIDA-16855-1; R01DA016855 (NIH); R01-16855-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Substance Abuse
Keywords: Contingency management; substance abuse treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management — Rewards (prizes) for abstinence

SUMMARY:
The purpose of this study is to train therapists to administer contingency management (CM). This project will train up to 42 community-based treatment providers about the rationale for and the specifics of administering CM. Initial training will occur in 2-day workshops, followed by weekly supervision in delivery of CM with test cases. We expect that the majority of therapists will achieve high levels of competence and adherence in administering CM treatment within 3-5 test cases, as measured by ratings of audiotapes. To examine the efficacy of CM, each therapist who achieves adherence and competence in delivering CM will administer standard treatment alone or standard treatment plus CM to substance-abusing outpatients. In the CM condition, patients will have the opportunity to win prizes for submission of negative samples, and the treatment will be in effect for 12 weeks. In total, up to 200 patients will be randomly assigned to one of the two conditions. A research evaluator will conduct follow-up assessments, scheduled for 3, 6 and 9 months after treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

Therapists who volunteer must have:

* at least one-year experience treating substance abusers, and at least 6 months employment at that center
* must commit to being available for both the workshop and individual training
* must be willing to allow random assignment of their patients to CM and non-CM treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
urinalysis results | baseline and at each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States